CLINICAL TRIAL: NCT00006128
Title: Study of Neurobehavioral Outcome in Children or Adolescents With Closed Head Injuries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Other Study IDs: 199/15289; BCM-H4373
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Head Injuries, Closed
Keywords: neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Head Injuries, Closed; Neurologic Manifestations; Mental Disorders; Rare Diseases

SUMMARY:
OBJECTIVES: I. Determine the relationship of closed head injury (CHI) severity, focal brain lesions, and the age at injury to the development of working memory, inhibition, and metacognitive skills in children or adolescents with CHI of varying severity.

II. Assess the development of working memory, inhibition, and metacognitive skills in relation to discourse functions, scholastic achievement, and adaptive behavior in these patients.

III. Determine the relationship between impaired inhibition, metacognitive skills, and the emergence of psychiatric disorder in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a multicenter study. Patients are assigned to one of two study groups based on when the closed head injury (CHI) occurred.

Study I (CHI that occurred at least 3 years ago): Patients undergo standardized and computer based testing of cognition, attention, planning ability, organizational ability, memory, fine motor functioning, reading and math skills, language, and behavioral and emotional functioning on day 1. Patients then undergo brain magnetic resonance imaging (MRI) on the same day. While each patient undergoes testing, the patient's parent/guardian answers interview questions regarding the patient's functional and emotional status since the injury, and the family's functional status, exposure to stressful events, and psychiatric history. Prior to the visit, a questionnaire regarding classroom behaviors, such as ability to focus in school and perform class work, is mailed to each patient's teacher.

Study II (recently diagnosed CHI): Patients undergo neurobehavioral and psychological testing as in study I once during hospitalization or soon after discharge, and then at 3, 6, 12, and 24 months. Patients undergo brain MRI at 3 months. While each patient undergoes testing, the patient's parent/guardian answers interview questions as in study I. Prior to each visit, the same questionnaire as in study I is mailed to each patient's teacher.

Both studies: A brief written summary of the patient's test results may be provided to the patient, parent/guardian, school, pediatrician, or other professional at the request of the patient and parent/guardian.

ELIGIBILITY:
* Study I: Closed head injury (CHI) that occurred at least 3 years ago
* Study II: Recently diagnosed CHI
* Both studies: Eligible if CHI resulted from acceleration, deceleration, or impact by a blunt object (e.g., motor vehicle accidents, pedestrian-vehicular injury, falls, assault except child abuse by caregiver) Preinjury emotional/behavioral problems allowed except mental retardation, autism, schizophrenia, or pervasive developmental disorder that would confound evaluation of cognitive function

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 374
Dates: Start 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S. Levin, Study Chair — Baylor College of Medicine
Locations (5):
- United States (4):
  - University of California San Diego Cancer Center, La Jolla, California
  - Callier Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas- Houston Medical School, Houston, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada